CLINICAL TRIAL: NCT03013270
Title: Aerobic, Resistance, Inspiratory Training Outcomes in Heart Failure. The ARISTOS-HF Trial: a Prospective Randomized Multicenter Trial
Brief Title: Aerobic, Resistance, Inspiratory Training Outcomes in Heart Failure
Acronym: ARISTOS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onassis Cardiac Surgery Centre (Other)
Collaborators: Asklepieion Voulas General Hospital (Other Government); National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Laoutaris Ioannis, PhD FESC, Onassis Cardiac Surgery Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARISTOS-HF
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: Rehabilitation; Exercise; Training
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ARIS group (Experimental): Aerobic-Resistance-Inspiratory
  Interventions: Other: Aerobic-Resistance-Inspiratory
- AT/RT group (Active Comparator): Aerobic-Resistance
  Interventions: Other: Aerobic-Resistance
- AT/IMT group (Active Comparator): Aerobic-Inspiratory
  Interventions: Other: Aerobic-Inspiratory
- AT group (Active Comparator): Aerobic Training
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Other: Aerobic-Resistance-Inspiratory — Patients will be submitted to a 12 week, 3 times/week, continuous aerobic (e.g. bike) training programme at an intensity of 60-80% max HR (or peakVO2) for 30 min combined with resistance training at an intensity of 50% of 1 Repetition Maximum (1RM) for quads training and upper limb exercises (elbow flex/shoulder flex/abd) using dumbbells (1-2 kg) (12-15 reps/3sets) for 10 min, combined also with inspiratory muscle training with a flow-resistive loading system at an intensity of 60% of maximal inspiratory pressure/sustained maximal inspiratory pressure (PImax/SPImax) for 20 min (Aerobic (30min) + Resistance (10min) + Inspiratory (20min) = 60 min)
  Arms: ARIS group
Other: Aerobic-Resistance — Patients will be submitted to a 12 week, 3 times/week, continuous aerobic (e.g. bike) training programme at an intensity of 60-80% max HR (or peakVO2) for 30 min combined with resistance training at an intensity of 50% of 1RM for quads training, pectoralis m, serratus anterior m, and latissimus dorsi m and upper limb exercises (elbow flex/shoulder flex/abd) using dumbbells (1-2 kg) (12-15 reps/3sets).
  (Aerobic (30min) + Resistance (30min) = 60 min)
  Arms: AT/RT group
Other: Aerobic-Inspiratory — Patients will be submitted to a 12 week, 3 times/week, continuous aerobic (e.g. bike) training programme at an intensity of 60-80% max HR (or peakVO2) for 30 min combined with inspiratory muscle training with a flow-resistive loading system at an intensity of 60% of maximal inspiratory pressure/sustained maximal inspiratory pressure (PImax/SPImax) for 30min (Aerobic (30min) + Inspiratory (30min) = 60 min)
  Arms: AT/IMT group
Other: Aerobic Training — Patients will be submitted to a 12 week, 3 times/week continuous aerobic (e.g. bike) training programme at an intensity of 60-80% max HR (or peakVO2) for 30 min combined with callisthenics progressing to treadmill or bike (at the same intensity) for 30 min (Aerobic training = 60 min)
  Arms: AT group

SUMMARY:
This study investigates the effects of aerobic, resistance, inspiratory training modalities outcomes in functional capacity and quality of life of heart failure (HF) patients, aiming for the 'optimum' (greek, αριστος=aristos) training program for HF patients.

DETAILED DESCRIPTION:
Heart failure is a clinical syndrome characterized by symptoms of dyspnea, exercise intolerance and decreased quality of life. A weakness in both inspiratory and peripheral muscles is also reported. Aerobic training (AT) improves the functional status of HF patients (level of evidence IA). Additional benefits of inspiratory muscle training (IMT) and/or resistance training (RT) when combined with aerobic training (AT) in HF symptoms have also been found.

Four exercise groups will be studied in order to identify the optimum exercise program I. Aerobic-Resistance-Inspiratory training (ARIS) group II. Aerobic Training-Resistance Training (AT/RT) group III. Aerobic training-Inspiratory Muscle Training (AT/IMT) group IV. Aerobic Training (AT) group

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (from New York Heart Association (NYHA) functional class II to NYHA III)
* Left ventricular ejection fraction below or equal to 35%

Exclusion Criteria:

* Uncontrolled arrhythmia
* Pulmonary oedema or pulmonary congestion in the last 30 days
* Cognitive, neurological or orthopaedic limitations
* Respiratory infection during 30 days before the start of the study
* Pulmonary limitations (e.g COPD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09; Primary Completion 2019-08 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
change in peak oxygen consumption (peakVO2, in ml/kg/min) using cardiopulmonary exercise testing (Medgraphics CPX/MAX, Medical Graphics Corp.,St. Paul, MN, USA, ZAN 600, ZAN Messgera¨te GmbH, Germany) | Before and after 12 weeks
  evaluation of maximal exercise capacity
change in left ventricular dimension (mm) using resting 2-dimensional echocardiography (Ultrasound Vivid 7 or 6, General Electric Healthcare, Fairfield, CT, USA) with the Teichholz method | Before and after 12 weeks
  evaluation of cardiac structure (LVEDD, LVESD in mm)

SECONDARY OUTCOMES:
change in walking distance using the 6-minute walking test (6MWT) | Before and after 12 weeks
  evaluation of submaximal exercise capacity
change in quality of Life using the Minnesota Living with Heart Failure questionnaire | Before and after 12 weeks
  evaluation of life quality
Preference Program Survey | After 12 weeks
  Questionnaire to evaluate exercise program preference (most enjoyed program) using a scale from 1 (=Very Little) to 5 (=Excellent)
change in left ventricular ejection fraction, echocardiography (Ultrasound Vivid 7 or 6, General Electric Healthcare, Fairfield, CT, USA) with the biplane Simpson' s method | Before and after 12 weeks
  evaluation of LVEF%

OTHER OUTCOMES:
Change in dyspnoea using the Borg scale (0-10) at the end of exercise testing | Before and after 12 weeks
  evaluation of dyspnea
Change in maximal inspiratory pressure (PImax in cmH2O) using an electronic pressure manometer with computer software (TRAINAIR®, Project Electronics Ltd, London, UK). | Before and after 12 weeks
  evaluation of inspiratory muscle strength
Change in inspiratory work capacity (sustained maximal inspiratory pressure (SPImax in cmH2O/s) using an electronic pressure manometer with computer software (TRAINAIR®, Project Electronics Ltd, London, UK). | Before and after 12 weeks
  evaluation of an inspiratory muscle endurance index
Change in skeletal muscle strength will be evaluated using the quadriceps 1 repetition maximum (1RM) | Before and after 12 weeks
  evaluation of skeletal muscle strength
Change in skeletal muscle endurance will be evaluated using the quadriceps muscle endurance with the product: 50%1Repetition Maximum x max number of reps | Before and after 12 weeks
  evaluation of skeletal muscle endurance
Morbidity Records | 6 months and 12 months after completion of Exercise Programs
  Evaluate Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Stamatis Adamopoulos, MD, Study Chair — Onassis Cardiac Surgery Center
Locations (3):
- Greece (2):
  - Onassis Cardiac Surgery Center, Athens, Attica
  - Asklepieion Voulas General Hospital, Voula, Attica
- Telecardiology Center, Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laoutaris ID, Adamopoulos S, Manginas A, Panagiotakos DB, Kallistratos MS, Doulaptsis C, Kouloubinis A, Voudris V, Pavlides G, Cokkinos DV, Dritsas A. Benefits of combined aerobic/resistance/inspiratory training in patients with chronic heart failure. A complete exercise model? A prospective randomised study. Int J Cardiol. 2013 Sep 1;167(5):1967-72. doi: 10.1016/j.ijcard.2012.05.019. Epub 2012 May 31. PMID 22658571
- [Background] Adamopoulos S, Schmid JP, Dendale P, Poerschke D, Hansen D, Dritsas A, Kouloubinis A, Alders T, Gkouziouta A, Reyckers I, Vartela V, Plessas N, Doulaptsis C, Saner H, Laoutaris ID. Combined aerobic/inspiratory muscle training vs. aerobic training in patients with chronic heart failure: The Vent-HeFT trial: a European prospective multicentre randomized trial. Eur J Heart Fail. 2014 May;16(5):574-82. doi: 10.1002/ejhf.70. Epub 2014 Mar 14. PMID 24634346
- [Background] Beckers PJ, Denollet J, Possemiers NM, Wuyts FL, Vrints CJ, Conraads VM. Combined endurance-resistance training vs. endurance training in patients with chronic heart failure: a prospective randomized study. Eur Heart J. 2008 Aug;29(15):1858-66. doi: 10.1093/eurheartj/ehn222. Epub 2008 May 30. PMID 18515805
- [Background] Smart NA. How do cardiorespiratory fitness improvements vary with physical training modality in heart failure patients? A quantitative guide. Exp Clin Cardiol. 2013 Winter;18(1):e21-5. PMID 24294043
- [Derived] Laoutaris ID, Piotrowicz E, Kallistratos MS, Dritsas A, Dimaki N, Miliopoulos D, Andriopoulou M, Manolis AJ, Volterrani M, Piepoli MF, Coats AJS, Adamopoulos S; ARISTOS-HF trial (Aerobic, Resistance, InSpiratory Training OutcomeS in Heart Failure) Investigators. Combined aerobic/resistance/inspiratory muscle training as the 'optimum' exercise programme for patients with chronic heart failure: ARISTOS-HF randomized clinical trial. Eur J Prev Cardiol. 2021 Dec 29;28(15):1626-1635. doi: 10.1093/eurjpc/zwaa091. PMID 33624071